CLINICAL TRIAL: NCT00140023
Title: A Multi-center, Open Label Study to Evaluate the Efficacy and Safety of Azithromycin Microspheres in Subjects Identified as Having Low Risk Community Acquired Pneumonia (CAP)
Brief Title: Azithromycin Microspheres in Patients With Low Risk Community Acquired Pneumonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0661149
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-05

CONDITIONS: Community-Acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia

INTERVENTIONS:
Drug: Azithromycin microspheres 2.0 single dose

SUMMARY:
The study will assess the clinical efficacy at Day 14-21 (Test of Cure), 14-21 days after starting the study drug; those subjects from whom a baseline pathogen is identified will also be assessed for bacteriologic response. All subjects who receive 1 dose of study medication will be assessed for safety.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years age or older, for whom oral, outpatient therapy is indicated.
* Diagnosis of CAP as manifested by at least 3 or more of the following:
* cough, pleuritic chest pain, fever (temperature of >37.8 C to <40 C), auscultatory findings on pulmonary examination of rales and/or evidence of pulmonary consolidation, dyspnea, tachypnea, laboratory results of elevated total peripheral white blood count (WBC> 10,000/mm3 or greater than 15% immature neutrophils (bands)

Exclusion Criteria:

* Known or suspected hypersensitivity or intolerance to azithromycin or other macrolides.
* Previously diagnosed disease(s) of immune function, including: subjects with baseline absolute neutrophil count < 1,000/mm3, HIV positive subjects with CD4 count < 200 cells/mm3, any immunoglobin or neutrophil disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2005-09; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the clinical efficacy of 2.0 g single dose of azithromycin microspheres in Low Risk CAP.

SECONDARY OUTCOMES:
To assess bacteriological efficacy of 2.0 g single dose of azithromycin microspheres. To assess the safety and tolerability of 2.0 g single dose of azithromycin microspheres.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- Philippines (5):
  - Pfizer Investigational Site, Manila, National Capital Region
  - Pfizer Investigational Site, City of Muntinlupa
  - Pfizer Investigational Site, Mandaluyong
  - Pfizer Investigational Site, Manila
  - Pfizer Investigational Site, Quezon City

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661149&StudyName=Azithromycin+Microspheres+in+Patients+with+Low+Risk+Community+Acquired+Pneumonia+